CLINICAL TRIAL: NCT00213525
Title: Genesis of Scleroderma: Role of Environmental Factors in 100 Patients With Scleroderma and 300 Healthy Controls
Brief Title: Genesis of Scleroderma: Role of Environmental Factors in 100 Patients With Scleroderma and 300 Controls
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2002/039/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients With Scleroderma: Assessments of questionnary for environmental factors research
  Interventions: Other: Questionnary for environmental factors research
- Healthy Controls: Assessments of questionnary for environmental factors research
  Interventions: Other: Questionnary for environmental factors research

INTERVENTIONS:
Other: Questionnary for environmental factors research — Questionnary for environmental factors research

SUMMARY:
Scleroderma is an autoimmune disease of unknown origin. Recently, the role of environmental factors, and particularly toxic drug exposure, in the genesis of scleroderma has been suggested.

This prompted us to conduct this prospective, case-control, multicentric study, including 2 groups of subjects:

* 100 patients with scleroderma
* 300 sex- and age-matched healthy controls. The aim of our study is to determine whether exposure to toxics is higher in patients with scleroderma compared with healthy controls.

DETAILED DESCRIPTION:
The data of patients with scleroderma and healthy controls will be compared regarding:

* a standardized questionnaire about "cursus laboris" at initial inclusion
* a search for toxics in blood, urine and hair: at initial exvaluation, 6 month and 2 year-follow-up

ELIGIBILITY:
Inclusion Criteria:

* patients with scleroderma with:

  * age range : 18 to 76 years
  * written consent

Exclusion Criteria:

* patients with other connective-tissue disorders
* pregnant women
* patients with psychiatric conditions
* unwritten consent

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 Patients With Scleroderma and 300 Healthy Controls
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2004-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Identification of environmental factor | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle MARIE, MD, PhD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, Rouen Cedex, France